CLINICAL TRIAL: NCT03702790
Title: Comparison of Clinical Impact in the Management of Patients With Spinal Pain Being Evaluated With Conventional SPECT Reconstruction vs. xSPECT
Brief Title: Comparison of Standard SPECT vs xSPECT Reconstruction in the Clinical Management of Patients With Spinal Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Principal Investigator, Jackson W Kiser, Medical Director Molecular Imaging, Carilion Clinic
Other Study IDs: 2585
Record Dates: First submitted 2018-10-04; First posted 2018-10-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Back pain SPECT evaluation: Patients with poorly localized back pain being imaged for clinical decision making

SUMMARY:
SPECT-CT is evolving into an integral part of patient management in those having back pain. It can supplement other types of imaging like MRI by providing physiologic information about the type and location of various disease processes. This information can help guide therapy to the most active sites of disease which MRI and CT cannot do as anatomic imaging modalities. The nuclear department has two cameras that are capable of performing SPECT-CT, an Optima manufactured by GE and a Symbia Intevo Bold manufactured by Siemens. The Optima uses the Volumetrix Evolution algorithm to reconstruct SPECT data that does not incorporate the CT data into these reconstructions. The Bold, on the other hand, has a proprietary reconstruction algorithm called xSPECT which does use the CT data to extract a zone map to better delineate tissue boundaries. In this study, the investigators hope to compare images using the standard and proprietary algorithms to determine if these provide equal or different levels of image interpretation confidence by the reader as well as changes in clinical management.

DETAILED DESCRIPTION:
Study objectives are: 1. Compare image quality between the Optima and Intevo as primary objective and 2.Does one device produce images that are more impactful on clinical management as a secondary objective.

The investigators have used both the Optima and Bold in their clinical practice for the evaluation of back pain in patients referred from sports medicine physicians and orthopedic spine surgeons. The two scanners and respective reconstruction algorithm software create distinctly different image sets. The investigators would like to do side by side comparison to determine if one device produces images of greater clinical value than the other.When patient is referred for a SPECT-CT scan for back pain, a standard injection of approximately 25mCi of MDP will be given. The patient will be then be randomly assigned to be scanned to either the Optima or the Intevo to be followed by scan on the other of the 2 scanners. Patients will be randomized as to the sequence of which scanner is used first or second so as to eliminate any potential bias that might occur due to variable uptake time of the radioisotope.

When scans are completed, images will be reviewed on PACS display and comparison will be made. Input as to the clinical impact of the images will also be assessed by the referring physicians to determine if one of the two scanners has superiority.

From the time of injection to the completion of both scans will be approximately 5 hours including a standard 3 hour uptake time after injection of the radioisotope. The scans will all be done on the same day with no return visits necessary. The interpreting radiologist will be blinded as to which scanner produced the images. Similarly, the referring physician will also be blinded when reviewing the images and determining patient management.The ordered exam is the standard of care and no ongoing treatments/therapies will be interrupted.

Study does not involve administering a therapy that would or would not be ultimately prescribed by the referring physician. Only exclusion criteria would be a known allergy to MDP used as the injected isotope. Pregnancy and claustrophobia that would prevent the patient from tolerating the SPECT-CT device would also be contraindications. The device is not experimental; it is an ongoing part of patient evaluation for back pain. The study wants to compare the impact of images using two separate reconstruction algorithms to determine superiority if present in the setting of clinical practice.

There is a very low risk of additional radiation exposure from the second low dose CT as part of the second SPECT-CT scan. Estimated additional exposure beyond dose administered for standard prescribed imaging protocol is approximately 1mSv or less. ALARA principles will be used as with all patients to use only as much dose as necessary to generate images.

ELIGIBILITY:
Inclusion Criteria:

* Poorly localized back pain in search for guided therapy

Exclusion Criteria:

* Allergy to MDP, radioisotope used for the examination. Patient limitations may include claustrophobia or inability to complete scan due to pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population are patients with back pain which cannot be definitively localized with other imaging procedures such as x-ray, CT or MRI
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Measure any change in management in patients with back pain based on results of two different SPECT reconstruction algorithms using a qualitative visual measure. | 1 year
  GE Optima vs Siemens Intevo

CONTACTS AND LOCATIONS:
Overall Officials: Jackson W Kiser, MD, Principal Investigator — Carilion Clinic
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Will discuss the results and outcomes of the study and present the data in the medical literature